CLINICAL TRIAL: NCT06807385
Title: Investigation of the Effect of the Reaction Training on Reaction Time, Anticipatory Postural Adjustment, and Balance in Parkinson's Disease
Brief Title: The Effect of the Reaction Training in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Mustafa Can Salamci, MSc, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-925
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Parkinson' Disease
Keywords: balance; reaction time; postural adjustments
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reaction Training Group (Experimental): In this group, we will use a reaction training and measurement system (Blazepod) for visual stimuli reaction training. Each exercise duration will be three minutes. The experimental group will apply reaction training two times a week for eight weeks. Each session will complet in 60 minutes.
  Interventions: Other: Reaction Training
- Control Group (Active Comparator): The exercises used in reaction training will be applied as in conventional training without visual aids. The difficulty of the exercise will be increased by changing the support surface and ground properties, taking the difficulty perceived by the individual as the criterion, as in reaction training.
  Interventions: Other: Conventional Exercises

INTERVENTIONS:
Other: Reaction Training — * The exercise list consists of 15 different exercises that aim to both shorten reaction time and improve stability with upper and lower extremity movements in different positions. In addition, the program includes both dual motor tasks and difficulties that require the physiotherapist to give the patient constantly changing motor tasks (tasks related to the color of the light to be touched, giving the command to read lights that are lit in different directions) and a second cognitive task.
  * Each station will be worked for 3 minutes, with at least 1 minute of rest between stations. Sessions will be planned by selecting the exercises in the exercise list for 60 minutes.
    * Appropriate modifications will be made to the station so that the difficulty of the exercise in the relevant station will be moderate (12-15 points) according to the Borg scale.
  Arms: Reaction Training Group
Other: Conventional Exercises — The exercises used in reaction training will be applied as in conventional training without reaction training system. The difficulty of the exercise will be increased by changing the support surface and ground properties, taking the difficulty perceived by the individual as the criterion, as in reaction training.
  The exercise list consists of 15 different exercises that aim to improve stability with upper and lower extremity movements in different positions. In addition, the program includes both dual motor tasks and difficulties that require the physiotherapist to give the patient constantly changing motor tasks and a second cognitive task. Each station will be worked for 3 minutes, with at least 1 minute of rest between stations. Sessions will be planned by selecting the exercises in the exercise list for 60 minutes. Appropriate modifications will be made to the station so that the difficulty of the exercise in the relevant station will be moderate (12-15 points for Borg Scale).
  Arms: Control Group

SUMMARY:
Parkinson's disease (PD) is one of the most common neurodegenerative diseases. Patients frequently experience decreased amplitude and speed of movements, balance, and gait problems. Although the basal ganglia have been the target neuroanatomical region for movement disorders in Parkinson's disease for many years, recent neuroscience studies have shown that the cerebellum also plays an important role in the disease and is an important alternative target for treatment applications. While medical applications are becoming current for this purpose, there is a significant deficiency in the literature in terms of physiotherapy applications. Reaction and dual task are activities that have been shown to naturally stimulate the cerebellum. The aim of this study is to examine the effects of combined exercise training, which includes dual skills and reaction activities that have been shown to stimulate the cerebellum in PD, on the reaction time, intuitive postural adjustments, and balance of PD. Our study is an original study that targets the cerebellum in PD with reaction training according to current neuroscience results, aims to contribute to the field of neuroscience and translational medicine, and has no previous example in the literature. This study will include patients diagnosed with idiopathic Parkinson's disease by a specialist physician. The PD patients included in the study will be randomly divided into two groups. The reaction group will be applied a combined reaction training program consisting of 15 exercises, including a light reaction measurement and an exercise system. The conventional group will be applied an exercise program consisting of only 15 exercises without reaction training. The patients included in the study will be subjected to reaction time, amplitude of intuitive postural adjustments, balance, and functional mobility assessments before and after the training. The light reaction measurement and exercise system will be applied for the measurement of reaction time of the volunteers, the static-dynamic balance assessment device for the assessment of intuitive postural adjustments and the static-dynamic balance assessment device for balance assessments, and the Timed Up and Go Test will be applied to assess functional mobility. At the end of the study, we aim to demonstrate the effect of combined exercise training targeting the cerebellum compared to conventional exercise training in Parkinson's patients, to create clinical outcomes for the inclusion of the cerebellum in more physiotherapy programs in Parkinson's disease, and to provide clinical outcomes for physiotherapists for a new exercise protocol, as well as making scientific contributions to the fields of translational medicine and neuroscience.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with "Parkinson's Disease" by a specialist neurologist according to the diagnostic criteria of the Movement Disorders Association
* Being between stages 1-3 according to the Hoehn and Yahr Staging
* Having additional neurological (migraine etc.), orthopedic (osteoarthritis etc.), cardiovascular (hypertension, benign arrhythmias etc.) diseases

Exclusion Criteria:

* Having a Standardized Mini-Mental Test score of >25
* Having a visual or hearing impairment that cannot be corrected with a device
* Having additional neurological (migraine etc.), orthopedic (osteoarthritis etc.), cardiovascular (hypertension, benign arrhythmias etc.) diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-11-06 (Actual)

PRIMARY OUTCOMES:
Postural Stability Assessment | Eight weeks
  Quantitative assessment of balance, allows the assessment of postural oscillations in different conditions such as two legs and one leg stance positions. For this purpose, a force platform (K-Force Platform, K-İnvent®) will be used for postural oscillations in different conditions. It will be done in two-leg stance with eyes open, in two-leg stance with eyes closed, and in one-leg stance. Each test will be performed 3 times.
Anticipatory Postural Adjustments Assessment | Eight weeks
  A force platform (K-Force Plate, K-İnvent) will be used to determine the amount of pressure center shift during the participants' stepping. Participants will be asked to stand on the force platform with their legs hip-width apart, in a posture as upright and stable as possible, and looking ahead at eye level. An audio stimulus will be used as a signal to start the movement. The measurement for the pressure center will be started 30 seconds before the signal to start the movement. Participants will be asked to stand in as upright and stable a position as possible for 30 seconds. At the end of 30 seconds, they will be asked to take the correct step first without waiting and as quickly as possible when they hear the audio stimulus. For the position analysis, the average and standard deviation of the positions in the 30-second standing position will be calculated.
Reaction Time Measurement | Eight weeks
  Measurement of reaction time will be done with the light reaction measurement and exercise system (Blazepod®) to be provided within the scope of the project for visual stimulus reaction training. There are two different concepts for reaction time: simple and choice. Simple reaction time is defined as the time between a single stimulus given and a single response. Choice reaction time is defined as the time between multiple stimuli given to the person and the appropriate response to the stimulus.
Movement Disorder Socity-Unified Parkinson's Disease Rating Scale | Eight weeks
  It was developed specifically for Parkinson's disease by Fahn and Elton in order to evaluate Parkinson's patients in terms of four clinical features. The scale, which includes a section for each clinical feature, consists of four sections in total. The first section consists of items that evaluate mental and emotional status (4 items); the second section includes items that evaluate daily living activities (13 items); the third section includes items that evaluate the severity of motor disorders (14 items); and the fourth section includes items that evaluate treatment-related complications (11 items). Scoring is done between zero and four in the total of 42 items in the scale, and a higher score indicates a more severe disorder. 0 points = Normal, 1 point = Slight, 2 points = Mild, 3 points = Moderate, 4 points = Severe. The validity and reliability of the Turkish version of the UPDRS were demonstrated in the study conducted by Akbostancı et al.

SECONDARY OUTCOMES:
Time Up and Go Test | Eight weeks
  The functional mobility of the patients will be assessed with the Timed Up and Go Test (TWG). In the test, the patient is asked to get up from the chair with the "walk" command, walk 3 m, turn around, and then sit back on the chair. The test is performed on a 3-meter flat surface.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lewis MM, Galley S, Johnson S, Stevenson J, Huang X, McKeown MJ. The role of the cerebellum in the pathophysiology of Parkinson's disease. Can J Neurol Sci. 2013 May;40(3):299-306. doi: 10.1017/s0317167100014232. PMID 23603164
- [Result] Gündüz, A. G., Otman, A. S., Köse, N., Bilgin, S., & Elibol, B. (2009). Parkinson hastalığında farklı denge ölçeklerinin karşılaştırılması. Fizyoterapi Rehabilitasyon, 20(1), 17-24.
- [Result] Gao L, Zhang J, Hou Y, Hallett M, Chan P, Wu T. The cerebellum in dual-task performance in Parkinson's disease. Sci Rep. 2017 Mar 30;7:45662. doi: 10.1038/srep45662. PMID 28358358
- [Result] Lupinacci NS, Rikli RE, Jones CJ, Ross D. Age and physical activity effects on reaction time and digit symbol substitution performance in cognitively active adults. Res Q Exerc Sport. 1993 Jun;64(2):144-50. doi: 10.1080/02701367.1993.10608791. PMID 8341837
- [Result] Akbostanci MC, Bayram E, Yilmaz V, Rzayev S, Ozkan S, Tokcaer AB, Saka E, Durmaz Celik FN, Barut BO, Tufekcioglu Z, Acarer A, Balaban H, Erer S, Dogu O, Kibaroglu S, Aydin N, Hanagasi H, Elibol B, Emre M, Stebbins GT, Goetz CG. Turkish Standardization of Movement Disorders Society Unified Parkinson's Disease Rating Scale and Unified Dyskinesia Rating Scale. Mov Disord Clin Pract. 2017 Nov 16;5(1):54-59. doi: 10.1002/mdc3.12556. eCollection 2018 Jan-Feb. PMID 30363359